CLINICAL TRIAL: NCT03906058
Title: Open-Label, Phase Ⅱ Study of Anlotinib Treatment in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma After Failure of no Less Than Second-line Chemotherapy or Targeted Therapy
Brief Title: Anlotinib in Recurrent or Metastatic Nasopharyngeal Carcinoma Patients After Failure of no Less Than Second-line Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2018-167
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib (Experimental)
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — All patients enrolled in the study will accept anlotinib treatment as a palliative treatment .

SUMMARY:
The purpose of this single arm, phase Ⅱ clinical trial is to evaluate the efficacy and safety of Anlotinib Treatment in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma after failure of no less than second-line chemotherapy or targeted therapy

ELIGIBILITY:
Inclusion Criteria:

* biopsy proved nasopharyngeal carcinoma;
* stage IVB according to American Joint Committee on Cancer(AJCC) edition VIII, or recurrent disease after chemotherapy and/or radiotherapy;
* 18 years or older; without other malignancy;
* proper functioning of the major organs.

Exclusion Criteria:

* allergic to anlotinib;
* female within gestation period or lactation;
* patients received drug of other clinical trial within 4 weeks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
disease control rate | 30 months
  disease control rate

SECONDARY OUTCOMES:
overall response rate | 30 months
  overall response rate
progression-free survival | 30 months
  progression-free survival
overall survival | 30 months
  overall survival
duration of response | 30 months
  duration of response

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Fang Y, Su N, Zou Q, Cao Y, Xia Y, Tang L, Tian X, Liu P, Cai Q. Anlotinib as a third-line or further treatment for recurrent or metastatic nasopharyngeal carcinoma: a single-arm, phase 2 clinical trial. BMC Med. 2023 Nov 7;21(1):423. doi: 10.1186/s12916-023-03140-x. PMID 37936166